CLINICAL TRIAL: NCT01620814
Title: Comparison of Intravaginal Misoprostol and Dinoprostol for the Purpose of Cervical Ripening Before Diagnostic Hysteroscopy in the Women at the Reproductive Age:RANDOMİSED,CONTROLLED PROSPECTİVE TRİAL
Brief Title: Intravaginal Misoprostol Versus Dinoprostone Before Diagnostik Hysteroscopy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Principal Investigator, Esra Tonguc, Assoc.Prof, Zekai Tahir Burak Women's Health Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-31
Record Dates: First submitted 2012-06-07; First posted 2012-06-15 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Cervical Ripening
Keywords: misoprostol; dinoprostone; cervical ripening; diagnostic hysteroscopy
MeSH Terms: interventions — Dinoprostone; Misoprostol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dinoprostone and misoprostol (Experimental): For the purpose of cervical ripening none procedure will be performed to Group 1, while vaginal misoprostole of 200 mg and vaginal dinoprostone will be applied to Group 2 and 3, respectively. While misoprostol will be implanted 3 hours before procedure, but dinoprostone will be implanted 6 hours before procedure. Before drug implantation for determination of the cervical insufficiency and measure of the cervical canal's opening, bougies will be applied toward to back from 8 no- hegar bougie.
  After drugs administration, cervical canal will be again evaluated with above mentioned way by bougie before hysteroscopy
  Interventions: Drug: Dinoprostone; Drug: misoprostol
- Misoprostol and control (Experimental): For the purpose of cervical ripening none procedure will be performed to Group 1, while vaginal misoprostole of 200 mg and vaginal dinoprostone will be applied to Group 2 and 3, respectively. While misoprostol will be implanted 3 hours before procedure, but dinoprostone will be implanted 6 hours before procedure. Before drug implantation for determination of the cervical insufficiency and measure of the cervical canal's opening, bougies will be applied toward to back from 8 no- hegar bougie.
  Interventions: Drug: misoprostol; Drug: control
- dinoprostone and control (Experimental): For the purpose of cervical ripening none procedure will be performed to Group 1, while vaginal misoprostole of 200 mg and vaginal dinoprostone will be applied to Group 2 and 3, respectively. While misoprostol will be implanted 3 hours before procedure, but dinoprostone will be implanted 6 hours before procedure. Before drug implantation for determination of the cervical insufficiency and measure of the cervical canal's opening, bougies will be applied toward to back from 8 no- hegar bougie.
  Interventions: Drug: Dinoprostone; Drug: control

INTERVENTIONS:
Drug: Dinoprostone
  Other Names: group 3
  Arms: Dinoprostone and misoprostol; dinoprostone and control
Drug: misoprostol
  Other Names: group 2
  Arms: Dinoprostone and misoprostol; Misoprostol and control
Drug: control
  Other Names: group 1
  Arms: Misoprostol and control; dinoprostone and control

SUMMARY:
Comparison of intravaginal misoprostol and dinoprostol for the purpose of cervical ripening before diagnostic hysteroscopy in the women at the reproductive age:RANDOMİSED,CONTROLLED PROSPECTİVE TRİAL Objective. Comparison with one another and with control group of vaginal dinoprostol and misoprostol with for the purpose of cervical ripening before diagnostic hysteroscopy.

Population: It was planned for performing to 95 women who appealed to gynecology polyclinic and will be performed diagnostic hysteroscopy.

Methods: Eighty-six women who will be performed diagnostic hysteroscopy assigned as randomize to three groups. It was planned that none procedure will be applied to group 1 for cervical ripening, vaginal misoprostol and vaginal dinoprostone will be practiced to Groups 2 and 3, respectively.

DETAILED DESCRIPTION:
While diagnostic hysteroscopy allows panoramic view of the uterus cavity, operational hysteroscopy allows to minimal invasive approach in the intrauterine lesions. Most frequently complications of hysteroscopy are cervical rupture, hemorrhage, failure of passage formation and uterus perforation. These generally are related to cervix dilatation's difficulty. These complications can be minimized preoperatively by the cervical ripening.

Present clinic study will be performed on the patients who appealed to gynecology polyclinic of the Konya TRH by the reason of infertility and infertility polyclinic of Zekai Tahir Burak Women Health Education and Research Hospital were planned diagnostic hysteroscopy by intrauterine pathology prediagnosis.Women will be given information about study and written informed consent will be obtained Inclusion criteria: On the HSG,USG or SIS, women at the age of primary or secondary infertile reproductive suspected for intrauterine pathology, no contraindication for hysteroscopy and reproductive age Exclusion criteria: Women are with allergy against to prostaglandins, with diseases in which prostaglandin usage is contraindicated, pregnant, don't given approval, with cervical surgery history and cervical insufficiency.

Post randomization. For the purpose of cervical ripening none procedure will be performed to Group 1, while vaginal misoprostole of 200 mg and vaginal dinoprostone will be applied to Group 2 and 3, respectively. While misoprostol will be implanted 3 hours before procedure, but dinoprostone will be implanted 6 hours before procedure. Before drug implantation for determination of the cervical insufficiency and measure of the cervical canal's opening, bougies will be applied toward to back from 8 no- hegar bougie.

After drugs administration, cervical canal will be again evaluated with above mentioned way by bougie before hysteroscopy, patients whose cervixes were easily passed via 5.5 no-hegar bougie, haven't cervical dislocation requirement and then directly hysteroscopy will be applied to them. Other patients will be applied cervical dislocation up to 6 no- hegar bougie before hysteroscopy. These processes also will be applied to patients of the Group 1.

ELIGIBILITY:
Inclusion Criteria:

* on the HSG,USG or SIS,
* women at the age of primary or secondary infertile reproductive suspected for intrauterine pathology,
* no contraindication for hysteroscopy and reproductive age

Exclusion Criteria:

* women are with allergy against to prostaglandins,
* with diseases in which prostaglandin usage is contraindicated,
* pregnant,
* don't given approval,
* with cervical surgery history and cervical insufficiency.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-07; Primary Completion 2012-08 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
need for cervical dilatation | 2 Months
  In the all three groups, patients being necessary cervical dilatation will be determined and their rates will be calculated.
Duration of cervical dilatation | 2 Months
  In the patients being necessary cervical dilatation, elapsed time for dilatation will be calculated.

SECONDARY OUTCOMES:
Ease of dilatation | 2 Months
  For determination of dilatation's ease 5-point Likert scale will be used.
Dilatation complications | 2 Months
  Cervical ruptures, haemorrhagee, uterine perforation and false passage will be evaluated as complication.
Adverse effects | 2 Months
  Side effects developing due to drugs in the patients who are in the drug treated- group will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Zekai Tahir Burak Women Health Education Research Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Inal HA, Ozturk Inal ZH, Tonguc E, Var T. Comparison of vaginal misoprostol and dinoprostone for cervical ripening before diagnostic hysteroscopy in nulliparous women. Fertil Steril. 2015 May;103(5):1326-31. doi: 10.1016/j.fertnstert.2015.01.037. Epub 2015 Feb 21. PMID 25712577